CLINICAL TRIAL: NCT03093948
Title: Effect of Remote Ischemic Post-conditioning on Neurologic and Cardiac Recovery in Out-of-hospital Cardiac Arrest
Brief Title: Effect of Remote Ischemic Post-conditioning on Out-of-hospital Cardiac Arrest
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Overlap with other RCT
Sponsor: Chonnam National University Hospital (Other)
Responsible Party: Principal Investigator, ByungKook Lee, Associate professor, Chonnam National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CNUH-2017-051
Record Dates: First submitted 2017-03-17; First posted 2017-03-28 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Out-Of-Hospital Cardiac Arrest
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remote Ischemic post-conditioning (Experimental)
  Interventions: Procedure: Remote ischemic post-conditioning
- standard of care (No Intervention)

INTERVENTIONS:
Procedure: Remote ischemic post-conditioning — Remote ischemic post-conditioning will undergo in both thighs at the beginning of targeted temperature management. This will be done with noninvasive measurement of blood pressure, with cuffs inflated to 200 mmHg for four 5 min cycles and interrupted three times for 5 min with cuff deflation.
  Arms: Remote Ischemic post-conditioning

SUMMARY:
Ischemia-reperfusion leads to mitochondrial injury, ion-pump injury, cell membrane damage, cytotoxic edema, and excessive oxygen free radical formation, and eventually destroys cells. Cardiac arrest is an example of global ischemia; after spontaneous circulation is restored, ischemia-reperfusion injury develops in cardiac arrest survivors.

Remote ischemic postconditioning (RIPoC) involves the application of brief, reversible episodes of ischemia and reperfusion to a vascular bed or tissue, rendering remote tissues and organs resistant to ischemia-reperfusion injury. Accordingly, RIPoC has been suggested as adjunctive therapy to mitigate ischemia-reperfusion injury. RIPoC applied by repeated brief inflation-deflation of a blood pressure cuff protects against myocardial injury, and has been proven effective in acute myocardial infarction.

This study aims to perform a randomized controlled trial to determine whether RIPoC has a neuroprotective effect and aids in myocardial recovery in out-of-hospital cardiac arrest patients after restoration of spontaneous circulation.

Neuron-specific enolase (NSE) at 48 hours after restoration of spontaneous circulation will be measured as a primary outcome.

ELIGIBILITY:
Inclusion Criteria:

* Adult (19 years and older)
* comatose out-of-hospital cardiac arrest with sustained restoration of spontaneous circulation
* Undergoing targeted temperature management
* Time of enrollment ≤ 6hrs from restoration of spontaneous circulation
* cardiac arrest from medical cause (cardiac or other medical cause)

Exclusion Criteria:

* Pre-existing dementia, brain injury, or dependence on others (cerebral performance category scale greater than 3)
* Traumatic etiology for cardiac arrest
* Protected population (pregnant, prisoner)
* in-hospital cardiac arrest
* Known bleeding diathesis
* suspected or confirmed acute intracranial hemorrhage
* suspected or confirmed acute ischemic stroke
* Known limitations in therapy and do-not-resuscitate order
* known disease making 180-day survival unlikely
* >6 hours from restoration of spontaneous circulation to randomization
* cardiac arrest from asphyxia (hanging, foreign body airway obstruction), drowning, drug overdose, or electrocution
* peripheral vascular disease (Deep vein thrombosis, arteriosclerosis obliterans)
* systolic blood pressure < 80 mmHg in spite of fluid loading/vasopressor and/or inotropic medication

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2017-03-21 (Actual); Primary Completion 2019-10-21 (Actual); Study Completion 2019-10-21 (Actual)

PRIMARY OUTCOMES:
neuron specific enolase | at 48 hour after restoration of spontaneous circulation
  expressed in ng/ml

SECONDARY OUTCOMES:
change over troponin-I | at 24 hour and 48 hour after restoration of spontaneous circulation
  troponin-I will be expressed in ng/ml
change over creatinin kinase-MB | at 24 hour and 48 hour after restoration of spontaneous circulation
  CK-MB will be expressed in ng/ml
neurologic outcome | an average of 3 weeks after restoration of spontaneous circulation
  cerebral performance category scale 1, 2, 3, 4, 5

OTHER OUTCOMES:
microRNA | at 48 hour after restoration of spontaneous circulation
  only in patients with shockable rhythm
neurologic outcome | six month after cardiac arrest
  cerebral performance category scale 1, 2, 3, 4, 5

CONTACTS AND LOCATIONS:
Overall Officials: Byungkook Lee, M.D., Principal Investigator — Department of Emergency Medicine, Chonnam National University Hospital
Locations (1):
- Chonnam National University Hospital, Gwangju, South Korea

REFERENCES:
- [Result] McNally B, Robb R, Mehta M, Vellano K, Valderrama AL, Yoon PW, Sasson C, Crouch A, Perez AB, Merritt R, Kellermann A; Centers for Disease Control and Prevention. Out-of-hospital cardiac arrest surveillance --- Cardiac Arrest Registry to Enhance Survival (CARES), United States, October 1, 2005--December 31, 2010. MMWR Surveill Summ. 2011 Jul 29;60(8):1-19. PMID 21796098
- [Result] Roger VL, Go AS, Lloyd-Jones DM, Adams RJ, Berry JD, Brown TM, Carnethon MR, Dai S, de Simone G, Ford ES, Fox CS, Fullerton HJ, Gillespie C, Greenlund KJ, Hailpern SM, Heit JA, Ho PM, Howard VJ, Kissela BM, Kittner SJ, Lackland DT, Lichtman JH, Lisabeth LD, Makuc DM, Marcus GM, Marelli A, Matchar DB, McDermott MM, Meigs JB, Moy CS, Mozaffarian D, Mussolino ME, Nichol G, Paynter NP, Rosamond WD, Sorlie PD, Stafford RS, Turan TN, Turner MB, Wong ND, Wylie-Rosett J; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2011 update: a report from the American Heart Association. Circulation. 2011 Feb 1;123(4):e18-e209. doi: 10.1161/CIR.0b013e3182009701. Epub 2010 Dec 15. PMID 21160056
- [Result] Iliodromitis EK, Kyrzopoulos S, Paraskevaidis IA, Kolocassides KG, Adamopoulos S, Karavolias G, Kremastinos DT. Increased C reactive protein and cardiac enzyme levels after coronary stent implantation. Is there protection by remote ischaemic preconditioning? Heart. 2006 Dec;92(12):1821-6. doi: 10.1136/hrt.2006.089060. Epub 2006 Jul 19. PMID 16855045
- [Result] Hoole SP, Heck PM, Sharples L, Khan SN, Duehmke R, Densem CG, Clarke SC, Shapiro LM, Schofield PM, O'Sullivan M, Dutka DP. Cardiac Remote Ischemic Preconditioning in Coronary Stenting (CRISP Stent) Study: a prospective, randomized control trial. Circulation. 2009 Feb 17;119(6):820-7. doi: 10.1161/CIRCULATIONAHA.108.809723. Epub 2009 Feb 2. PMID 19188504
- [Result] Davies WR, Brown AJ, Watson W, McCormick LM, West NE, Dutka DP, Hoole SP. Remote ischemic preconditioning improves outcome at 6 years after elective percutaneous coronary intervention: the CRISP stent trial long-term follow-up. Circ Cardiovasc Interv. 2013 Jun;6(3):246-51. doi: 10.1161/CIRCINTERVENTIONS.112.000184. Epub 2013 May 21. PMID 23696599
- [Result] Ahmed RM, Mohamed el-HA, Ashraf M, Maithili S, Nabil F, Rami R, Mohamed TI. Effect of remote ischemic preconditioning on serum troponin T level following elective percutaneous coronary intervention. Catheter Cardiovasc Interv. 2013 Nov 1;82(5):E647-53. doi: 10.1002/ccd.24825. Epub 2013 Jun 18. PMID 23404916
- [Result] Prasad A, Gossl M, Hoyt J, Lennon RJ, Polk L, Simari R, Holmes DR Jr, Rihal CS, Lerman A. Remote ischemic preconditioning immediately before percutaneous coronary intervention does not impact myocardial necrosis, inflammatory response, and circulating endothelial progenitor cell counts: a single center randomized sham controlled trial. Catheter Cardiovasc Interv. 2013 May;81(6):930-6. doi: 10.1002/ccd.24443. Epub 2012 Nov 8. PMID 22517646
- [Result] Luo SJ, Zhou YJ, Shi DM, Ge HL, Wang JL, Liu RF. Remote ischemic preconditioning reduces myocardial injury in patients undergoing coronary stent implantation. Can J Cardiol. 2013 Sep;29(9):1084-9. doi: 10.1016/j.cjca.2012.11.022. Epub 2013 Feb 12. PMID 23414904
- [Result] Xu X, Zhou Y, Luo S, Zhang W, Zhao Y, Yu M, Ma Q, Gao F, Shen H, Zhang J. Effect of remote ischemic preconditioning in the elderly patients with coronary artery disease with diabetes mellitus undergoing elective drug-eluting stent implantation. Angiology. 2014 Sep;65(8):660-6. doi: 10.1177/0003319713507332. Epub 2013 Oct 24. PMID 24163121
- [Result] Zografos TA, Katritsis GD, Tsiafoutis I, Bourboulis N, Katsivas A, Katritsis DG. Effect of one-cycle remote ischemic preconditioning to reduce myocardial injury during percutaneous coronary intervention. Am J Cardiol. 2014 Jun 15;113(12):2013-7. doi: 10.1016/j.amjcard.2014.03.043. Epub 2014 Apr 1. PMID 24793669
- [Result] Munk K, Andersen NH, Schmidt MR, Nielsen SS, Terkelsen CJ, Sloth E, Botker HE, Nielsen TT, Poulsen SH. Remote Ischemic Conditioning in Patients With Myocardial Infarction Treated With Primary Angioplasty: Impact on Left Ventricular Function Assessed by Comprehensive Echocardiography and Gated Single-Photon Emission CT. Circ Cardiovasc Imaging. 2010 Nov;3(6):656-62. doi: 10.1161/CIRCIMAGING.110.957340. Epub 2010 Sep 8. PMID 20826592
- [Result] Rentoukas I, Giannopoulos G, Kaoukis A, Kossyvakis C, Raisakis K, Driva M, Panagopoulou V, Tsarouchas K, Vavetsi S, Pyrgakis V, Deftereos S. Cardioprotective role of remote ischemic periconditioning in primary percutaneous coronary intervention: enhancement by opioid action. JACC Cardiovasc Interv. 2010 Jan;3(1):49-55. doi: 10.1016/j.jcin.2009.10.015. PMID 20129568
- [Result] Crimi G, Pica S, Raineri C, Bramucci E, De Ferrari GM, Klersy C, Ferlini M, Marinoni B, Repetto A, Romeo M, Rosti V, Massa M, Raisaro A, Leonardi S, Rubartelli P, Oltrona Visconti L, Ferrario M. Remote ischemic post-conditioning of the lower limb during primary percutaneous coronary intervention safely reduces enzymatic infarct size in anterior myocardial infarction: a randomized controlled trial. JACC Cardiovasc Interv. 2013 Oct;6(10):1055-63. doi: 10.1016/j.jcin.2013.05.011. PMID 24156966
- [Result] Sloth AD, Schmidt MR, Munk K, Kharbanda RK, Redington AN, Schmidt M, Pedersen L, Sorensen HT, Botker HE; CONDI Investigators. Improved long-term clinical outcomes in patients with ST-elevation myocardial infarction undergoing remote ischaemic conditioning as an adjunct to primary percutaneous coronary intervention. Eur Heart J. 2014 Jan;35(3):168-75. doi: 10.1093/eurheartj/eht369. Epub 2013 Sep 12. PMID 24031025